CLINICAL TRIAL: NCT05696275
Title: Exercise-aided Caring System With Dual-mode Assessment Method Using ePRO and Wearables for Cancer-related Fatigue
Brief Title: Using Combine Walking and Elastic Band to Decrease Fatigue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Tsai-Wei Huang, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N202208012
Record Dates: First submitted 2022-11-16; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Cancer Related Fatigue
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise (Experimental): combine walking and elastic band exercise
  Interventions: Behavioral: exercise
- usual care (No Intervention): as usual care

INTERVENTIONS:
Behavioral: exercise — 20-30 minutes of walking and elastic band exercise per day
  Arms: exercise

SUMMARY:
This study is expected to propose an industry-university cooperation research case for the next two years. When cancer patients use ePRO to record subjective fatigue, and smart watches with 4G communication record objective fatigue, they will be given according to the patient's current degree of mild, moderate and severe fatigue. Suffer from 'exercise or activity' advice and lead the implementation of appropriate exercise advice. This study is expected to design aerobic + anaerobic exercise suitable for mild or moderate patients, and use the sensor of the smart watch to monitor the effect of exercise and fatigue. To sum up, the first-year plan is expected to use the established ePRO electronic records, combined with the LINE communication system, to integrate into a "cancer-related fatigue electronic registration and care system"; the second-year plan will integrate objective fatigue classifiers, Establish the exercise care option in the fatigue care system, and use the smart watch to establish a technology record function of the exercise process to help track the fatigue level of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. age 20 years old;
2. diagnosis of cancer;
3. can continuous wearing bracelet for 14 days or more

Exclusion Criteria:

1. Unclear and unable to answer the questionnaire；
2. Not able to walk；
3. platelet <50,000/mm3；
4. ANC 500/cumm

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-16 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
cancer fatigue--BFI | Change from Baseline post exercise 5 min
  severity of fatigue level; measurement tool: Brief Fatigue Index
cancer fatigue--BFI | Change from Baseline at 1 month.
  severity of fatigue level; measurement tool: Brief Fatigue Index

SECONDARY OUTCOMES:
Physical Activity assessment--IPAQ | Change from Baseline post exercise 5 min
  International Physical Activity Questionnaire (IPAQ), the questionnaire consists of seven questions regarding types of physical activity that constitute elements of everyday life. The questions refer to physical activity in the last seven days and concern the time spent sitting and walking as well as the time devoted to vigorous and moderate physical activity. Activities done for at least 10 min at a time are taken into account. This instrument is used to assess physical activity levels-according to the IPAQ scoring protocol, three levels are distinguished, i.e., low, moderate and high.
Physical Activity assessment--IPAQ | Change from Baseline at 1 month.
  International Physical Activity Questionnaire (IPAQ), the questionnaire consists of seven questions regarding types of physical activity that constitute elements of everyday life. The questions refer to physical activity in the last seven days and concern the time spent sitting and walking as well as the time devoted to vigorous and moderate physical activity. Activities done for at least 10 min at a time are taken into account. This instrument is used to assess physical activity levels-according to the IPAQ scoring protocol, three levels are distinguished, i.e., low, moderate and high.
Chinese version of the Edmonton Symptom Assessment System，C-ESAS | Change from Baseline post exercise 5 min
  The ESAS includes 11 symptoms: pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, sleep, well-being, shortness of breath, and other. It uses a 0-10 numerical scale: 0 shows the absence of a symptom, and 10 shows the worst experience of the symptom.
Chinese version of the Edmonton Symptom Assessment System，C-ESAS | Change from Baseline at 1 month.
  The ESAS includes 11 symptoms: pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, sleep, well-being, shortness of breath, and other. It uses a 0-10 numerical scale: 0 shows the absence of a symptom, and 10 shows the worst experience of the symptom.
Sleep quality--PSQI | Change from Baseline post exercise 5 min
  Pittsburgh Sleep Quality Index (PSQI) scores, is used to assess the quality of sleep of patients - with scores ranging from 0 to 21 - with lower scores indicating better sleep quality.
Sleep quality--PSQI | Change from Baseline at 1 month.
  Pittsburgh Sleep Quality Index (PSQI) scores, is used to assess the quality of sleep of patients - with scores ranging from 0 to 21 - with lower scores indicating better sleep quality.
Steps count | Change from Baseline post exercise 5 min
  more steps means good for ability
Steps count | Change from Baseline at 1 month.
  more steps means good for ability
walking distance | Change from Baseline post exercise 5 min
  Longer distances mean better movement
walking distance | Change from Baseline at 1 month.
  Longer distances mean better movement
strength ability | Change from Baseline post exercise 5 min
  Muscle strength is measured with a muscle strength meter, and an increase in value means an increase in muscle strength
strength ability | Change from Baseline at 1 month.
  Muscle strength is measured with a muscle strength meter, and an increase in value means an increase in muscle strength
Smart bracelet_Heart rate variability (HRV) | Continue wear bracelet five days to record HRV data.
  HRV is the physiological phenomenon of the variation in the time interval between consecutive heartbeats in milliseconds. A normal, healthy heart does not tick evenly like a metronome, but instead, when looking at the milliseconds between heartbeats, there is constant variation.

IPD SHARING:
Plan to Share IPD: No